CLINICAL TRIAL: NCT02110654
Title: Comparison of Daily Mometasone Furoate Nasal Spray Alone Versus a Combination With Montelukast for Treatment of Chronic Rhinosinusitis With Asthma After Functional Endoscopic Sinus Surgery: a 9-month Randomized, Open-label, Controlled Study
Brief Title: Comparison of Daily Mometasone Furoate Nasal Spray Alone Versus a Combination With Montelukast for Treatment of Chronic Rhinosinusitis With Asthma After Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jianbo Shi, Deputy director of ENT department, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20140329
Record Dates: First submitted 2014-03-31; First posted 2014-04-10 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Sinusitis; Nasal Polyps; Asthma
Keywords: chronic rhinosinusitis; asthma; montelukast; surgery; treatment outcomes
MeSH Terms: conditions — Sinusitis; Nasal Polyps; Asthma | interventions — montelukast; Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: There are two study groups listed as below.
  1. Montelukast 10mg once daily + Mometasone furoate nasal spray 100 µg/per nostril once daily for 6 months.
  2. Mometasone furoate nasal spray 100 µg/per nostril once daily for 6 months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mometasone furoate nasal spray (Active Comparator): mometasone furoate nasal spray,200ug qd, 6 months
  Interventions: Drug: Montelukast
- mometasone furoate nasal spray combined with montelukast (Experimental): montelukast tablet,10mg,qd + mometasone furoate nasal spray, 200ug qd,6 months
  Interventions: Drug: Montelukast; Drug: mometasone furoate nasal spray

INTERVENTIONS:
Drug: Montelukast
  Other Names: singulair
Drug: mometasone furoate nasal spray
  Other Names: nasonex
  Arms: mometasone furoate nasal spray combined with montelukast

SUMMARY:
1. objectives. To compare the efficacy and the safety of mometasone furoate nasal spray (MFNS; Nasonex 200μg, daily) alone versus a combination with montelukast (singulair 10mg, daily) in chronic rhinosinusitis (CRS) with asthma after functional endoscopic sinus surgery (FESS) for improvement the clinical control of CRS
2. the clinical hypotheses. The investigators hypothesize that postoperative combined montelukast and MFNS can better improve clinical control of CRS concomitant with asthma after FESS compared with MFNS alone.
3. study design This study is a 9-month randomized, open-label, controlled interventional study.

DETAILED DESCRIPTION:
1. Surgery plan

   * Pre-operation: Patients enrolled in the study will complete assessment and specimen collection on the first day, then followed by 1 week drug therapy with prednisone (30 mg once daily) and MFNS(200ug, once daily).
   * FESS: For patients with no surgical contraindications, FESS will be performed. Bilateral nasal cavities will be filled with swelling sponges postoperatively. The stuffing will be removed on postoperative day 2. The patients will be discharged on day 3 after surgery.
   * Other treatment: All patients will receive nasal irrigation (normal saline 500 mg twice daily) from postoperative day 3 until day 30. Asthma will be treated as the guidance of professors from the Department of Respiratory Medicine in the investigators hospital.
2. Drug treatment phase Three days after the surgery (FESS) described above, all patients will be assigned to the following two groups (30 patients each group) using random numbers generated by statistical software.

   * Experimental group: Montelukast (10mg, once daily) and MFNS (200μg, once daily) for 6 months
   * Control group: MFNS (200μg, once daily) for 6 months
3. Follow up After the 6-month drug treatment phase, there are still a 3-month follow-up. Totally, there are 5 visits after FESS surgery.

   * Visit 1: baseline
   * Visit 2： Day 31 post-FESS
   * Visit 3: Day 61 post-FESS
   * Visit 4: Day 91 post-FESS
   * Visit 5: Day 181 post-FESS
   * Visit 6: Day 271 post-FESS

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic rhinosinusitis according to European position paper of rhinosinusitis and nasal polyps 2007
2. Diagnosis of asthma based on Global initiative for asthma 2012
3. All patients should provide informed consent prior to the study and agree to follow-up appointments.

Exclusion Criteria:

1. Immunodeficiency diseases, history of head and/or facial trauma, cancer or organ transplant recipients.
2. Pregnancy or lactation.
3. Uncontrolled bronchial asthma.
4. Acute respiratory tract infection within one month before the study.
5. Use of leukotriene receptor antagonist within 3 months before the enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Decrease in Nasal symptome Visual Analogue Scale (VAS) | 9 months
  nasal symptoms include general symptom, congestion, rhinorrhea, olfactory loss and headache.

SECONDARY OUTCOMES:
Percentage of Participants with Decrease in nasal endoscopy score (Lund-Kennedy score) | 9 months
  Visit 1: baseline Visit 2：Day 31 post-FESS Visit 3: Day 61 post-FESS Visit 4: Day 91 post-FESS Visit 5: Day 181 post-FESS Visit 6: Day 271 post-FESS
Percentage of Participants with Decrease in sinus CT score (Lund-Mackay, scoring system) | 6 months
  baseline, 6 months post-FESS
Percentage of Participants with Increase in Asthma Control test (ACT) | 9 months
  Visit 1: baseline Visit 2：Day 31 post-FESS Visit 3: Day 61 post-FESS Visit 4: Day 91 post-FESS Visit 5: Day 181 post-FESS Visit 6: Day 271 post-FESS
Number of Participants with Serious and Non-Serious Adverse Events | 9 months
  Visit 1: baseline Visit 2：Day 31 post-FESS Visit 3: Day 61 post-FESS Visit 4: Day 91 post-FESS Visit 5: Day 181 post-FESS Visit 6: Day 271 post-FESS

CONTACTS AND LOCATIONS:
Overall Officials: jianbo shi, doctor, Study Director — Ent department, the first affiliated hospital, Sun Yat-sen University
Locations (1):
- the first affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hong H, Chen F, Sun Y, Yang Q, Gao W, Cao Y, Fan Y, Shi J, Li H. Nasal IL-25 predicts the response to oral corticosteroids in chronic rhinosinusitis with nasal polyps. J Allergy Clin Immunol. 2018 May;141(5):1890-1892. doi: 10.1016/j.jaci.2017.10.050. Epub 2018 Jan 11. No abstract available. PMID 29337030
- [Derived] Chen F, Hong H, Sun Y, Hu X, Zhang J, Xu G, Zhao W, Li H, Shi J. Nasal interleukin 25 as a novel biomarker for patients with chronic rhinosinusitis with nasal polyps and airway hypersensitiveness: A pilot study. Ann Allergy Asthma Immunol. 2017 Oct;119(4):310-316.e2. doi: 10.1016/j.anai.2017.07.012. Epub 2017 Sep 1. PMID 28870448